CLINICAL TRIAL: NCT06980896
Title: Exploratory Pathophysiological Study on the Association Between Physical Performance and Biomarkers of Oxidative Stress and Low-Grade Inflammation in Elderly Patients
Brief Title: Physical Activity Oxidative Stress and Inflammation With Ageing
Acronym: POXI-AGEING
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Société KONDREE (Unknown); Laboratoire PhyMedExp (Unknown); CHU de Liège, Pr Pincemail (Unknown)
Responsible Party: Principal Investigator, bp-prom-regl, Dr Guillaume Chapelet, Nantes University Hospital
Other Study IDs: RC24_0365
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Inflammation; Oxydative Stress; Sarcopenia; Older Patient; Ageing
Keywords: inflammation; oxydative stress; sarcopenia; older patient; ageing
MeSH Terms: conditions — Inflammation; Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- slightly frail elderly, but excludes those with marked weight loss, low BMI: In this study, participants will undergo scheduled assessments, including blood tests, physical performance evaluations, and nutritional intake monitoring. Participants will be excluded from the study if they meet any of the following conditions: significant weight loss, defined as a reduction of more than 5% in one month or more than 10% in six months, Body Mass Index (BMI) below 22 kg/m², lifestyle and medical conditions that could interfere with study outcomes (smoking, diabetes, active cancer or cancer treatment within the past five years, chronic inflammatory diseases, recent infections or inflammatory episodes within the past month, long-term corticosteroid therapy or corticosteroid use within the last month, use of antioxidant supplements (including vitamins C and E, zinc, or selenium) within the past three monthscorticosteroid use within the last month, use of antioxidant supplements (including vitamins C and E, zinc or selenium) within the past three months

SUMMARY:
Sarcopenia, an age-related decline in muscle function, are thought to be influenced by oxidative stress and low-grade inflammation, resulting in significant muscle mass reduction and altered physical performance. Indeed, oxidative stress and chronic inflammation in older adults are key factors contributing to metabolic protein disturbances, DNA mutations, and skeletal muscle decline during aging. Additionally, reduced food intake can lead to malnutrition, exacerbating muscle protein loss, oxidative stress and chronic inflammation.

Recent research has shown that a nutritional intervention, i.e. antioxidant supplementation (e.g., vitamins C, E, zinc, selenium) can reduce muscle damage in Facioscapulohumeral Dystrophy (FSHD) by correcting mitochondrial dysfunction and inflammation with a beneficial effect on physical performance and have led to the development of a personalized antioxidant supplementation model, supported by clinical trials (NCT02622438).

Although antioxidant supplementation appears beneficial for FSHD patients, its effects on age-related muscle decline remain unclear. This study aims to explore correlation between oxidative stress, inflammation, nutritional status and physical performance in older individuals. The findings will help establish the physiological basis for a potential antioxidant therapy for age-related muscle deterioration.

DETAILED DESCRIPTION:
The POXI-Ageing study aims to explore the relationship between oxidative stress, chronic inflammation, and muscle function in older individuals. The research hypothesizes that these biological factors contribute to muscle deterioration, commonly associated with aging, and may play a role in ageing conditions like sarcopenia. This prospective, exploratory, single-center, non-controlled study study will be conducted in CHU de Nantes (a French University Hospital in Nantes, France), and will included 30 participants (15 men and 15 women) at the Centre Ambulatoire Nantais de Gérontologie Clinique (CANGC), the geriatric outpatient clinic. The study is planned to run for a total of 17 months, divided into three key phases, a recruitment phase of 12 months, a follow-up Phase (up to 3 months), and a results/statistical analysis phase of 2 month.

In this study, participants will undergo scheduled assessments, including blood tests, physical performance evaluations, and nutritional intake monitoring. To participate in the study, individuals must meet the following conditions: (i) be aged between 70 and 90 years, (ii) have a scheduled blood test within two months, (iii) have a Clinical Frailty Score (CFS) of 4 or lower (indicating mild frailty). Participants will be excluded from the study if they meet any of the following conditions: significant weight loss, defined as a reduction of more than 5% in one month or more than 10% in six months, Body Mass Index (BMI) below 22 kg/m², lifestyle and medical conditions that could interfere with study outcomes (smoking, diabetes, active cancer or cancer treatment within the past five years, chronic inflammatory diseases, recent infections or inflammatory episodes within the past month, long-term corticosteroid therapy or corticosteroid use within the last month, use of antioxidant supplements (including vitamins C and E, zinc, or selenium) within the past three months.

Regarding g the cinlsuion process, and more in details, a presentation poster about the study will be placed in the waiting room of the outpatient clinic. Screening will be conducted during the patient's first visit to the day hospital at CANGC (V0), with an initial verification of inclusion and non-inclusion criteria. Only patients meeting these criteria and scheduled for other appointments/consultations at CANGC (up to 3 month), with a blood test indicated within the next two months, may be pre-included in the protocol. An oral explanation will be provided by the clinician during this V0 visit, along with the distribution of the information letter. Patients will have a reflection period and will be able to ask the doctor any questions if needed. Patients who express their willingness to participate and indicate their non-opposition to the study will be considered pre-included. They will then be contacted by phone approximately 20 days before visit V1, which corresponds to their median next routine care appointment, to remind them of the instructions to follow before the blood and urine sample collection. A re-evaluation of the inclusion and non-inclusion criteria will be conducted on the day of V1 before their official inclusion in the study. This step will precede the blood sampling, urine collection, and the specific physical tests and examinations required for the research.

The primary objective will be to describe and investigate correlations between oxidative stress biomarkers, inflammation biomarkers, and muscle strength in older patients. The primary outcome will be Vitamin C/Vitamin E ratio, Copper/Zinc ratio, Selenium levels, and muscle strength, measured using an hand grip strength test and a quadriceps isometric contraction strength test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 70 to 90, consulting the Nantes CHU CANGC (Bellier Hospital) and who has an indication for a blood test scheduled as part of routine care within 4 months according to the clinician.
* Clinical Frailty Scale (CFS) score less than or equal to 4 (i.e. threshold for identifying frail elderly people).

Exclusion Criteria:

* Opposition to participation in the study
* Indication for emergency blood sampling in the city
* Use of a wheelchair or with a proven disability
* Criteria for undernutrition: weight loss of more than 5% in the last month or more than 10% in the last 6 months and/or BMI strictly less than 22 kg/m2.
* Tobacco consumption
* Diabetes
* Any type of active and/or treated cancer less than 5 years old
* Chronic inflammation pathology
* Clinically significant infectious or inflammatory episode ended at least one month ago
* Long-term or last-month corticosteroid therapy
* Antioxidants or trace elements taken in the last 3 months
* Patient not affiliated to a Social Security system
* Patient deprived of liberty by judicial or administrative decision
* Patients under guardianship or trusteeship

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients consulting at the geriatric outpatient clinic in Nantes University Hospital (Nantes, France)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlations between VitC/VitE and Cu/Zn ratios, selenium, and muscle strength | 8 months
  Correlations between VitC/VitE and Cu/Zn ratios, selenium, and muscle strength assessed according to EWGSOP(2) recommendations: hand grip strength (in kg) measured using the Baseline® model 12-0286, and quadriceps strength (in kg, isometric contraction) measured using a testing bench coupled with Biopac exploitation software (MP SYSTEM, ACQKnowledge®: MP36 Pack BASIC with BSL4 Software).

SECONDARY OUTCOMES:
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and muscle strength in the included patients. | 8 months
  Correlations between the biomarkers listed below and muscle strength, as evaluated for the primary outcome according to EWGSOP(2) recommendations.
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and muscle power in the included patients. | 8 months
  Correlations between all biomarkers directly or indirectly involved in oxidative stress, cited in the primary outcome and in secondary outcome #1, and muscle power measured by the Five-Time Sit-to-Stand Test (FTSST) in seconds.
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and muscle mass in the included patients. | 8 months
  Correlations between all biomarkers directly or indirectly involved in oxidative stress, cited in the primary outcome and in secondary outcome #1, and appendicular skeletal muscle mass (ASM), assessed by segmental bioimpedance using the BIACORPUS RX 4004M and BODYCOMP software in kg for upper and lower limbs, as well as the ASM index (ASMI = ASM/height²).
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and physical performance in the included patients. | 8 months
  Correlations between all biomarkers directly or indirectly involved in oxidative stress, cited in the primary outcome and in secondary outcome #1, and physical performance assessed according to EWGSOP(2) recommendations: Timed Up and Go (TUG) in seconds and 4-meter walking speed in m/s.
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and inflammatory biomarkers in the included patients. | 8 months
  Correlations between all biomarkers directly or indirectly involved in oxidative stress, cited in the primary outcome and in secondary outcome #1, and inflammatory biomarkers, including:
  * HCYTOMAG-60K Panel: sCD40L, EGF, FGF-2, Flt-3 ligand, Fractalkine, G-CSF, GM-CSF, GRO, IFN-α2, IFN-γ, IL-1α, IL-1β, IL-1ra, IL-2, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12(p40), IL-12(p70), IL-13, IL-15, IL-17A, IP-10, MCP-1, MCP-3, MDC (CCL22), MIP-1α, MIP-1β, PDGF-AB/BB, RANTES, TGF-α, TNF-α, TNF-β, VEGF, Eotaxin/CCL11, PDGF-AA.
  * Human Aging Magnetic Bead Panel 1 - Metabolism Multiplex Assay: CTACK (skin chemokines), FGF-21, GDF-15, IL-6, IL-10, IL-18, Leptin.
  * Other markers: Fibrinogen, CRP.
Investigate correlations between biomarkers involved directly or indirectly in the oxidative stress process and the nutritional intake of the included patients. | 8 months
  Correlations between all biomarkers directly or indirectly involved in oxidative stress, cited in the primary outcome and in secondary outcome #1, and the following average nutritional intakes, estimated using GENI v9.6 software and the Phenol-Explorer database version 3.6 for polyphenols, based on a 3-day dietary record (2 non-consecutive weekdays and 1 weekend day), following the recommendations of the French National Institute for Prevention and Health Education (INPES)
Investigate correlations between inflammation-related biomarkers and muscle strength in the included patients. | 8 months
  Correlations between inflammation-related biomarkers (cited in secondary outcome #5) and muscle strength, as evaluated for the primary outcome.
Investigate correlations between inflammation-related biomarkers and muscle power in the included patients. | 8 months
  Correlations between inflammation-related biomarkers (cited in secondary outcome #5) and muscle power, as measured for secondary outcome #2.
Investigate correlations between inflammation-related biomarkers and muscle mass in the included patients. | 8 months
  Correlations between inflammation-related biomarkers (cited in secondary outcome #5) and appendicular skeletal muscle mass (ASM), as evaluated for secondary outcome #3.
Investigate correlations between inflammation-related biomarkers and physical performance in the included patients. | 8 months
  Correlations between inflammation-related biomarkers (cited in secondary outcome #5) and physical performance, as evaluated for secondary outcome #4.
Investigate correlations between inflammation-related biomarkers and the nutritional intake of the included patients. | 8 months
  Correlations between inflammation-related biomarkers (cited in secondary outcome #5) and average nutritional intake, as estimated for secondary outcome #6.
Investigate correlations between nutritional intake and physical performance in the included patients. | 8 months
  Correlations between estimated nutritional intake (secondary outcome #6) and physical performance (secondary outcome #4).
Investigate correlations between muscle mass and physical performance in the included patients. | 8 months
  Correlations between estimated nutritional intake (secondary outcome #6) and physical performance (secondary outcome #4).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Anthony Dylis, Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No